CLINICAL TRIAL: NCT01121042
Title: Double Blind, Placebo-Controlled, Randomised Investigation of Ondansetron in Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 145/10
Record Dates: First submitted 2010-05-09; First posted 2010-05-12 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Schizoaffective and Schizophreniform Disorders; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ondansetron (Active Comparator): Ondansetron oral capsule 8mg daily
  Interventions: Drug: Ondansetron
- Placebo (Placebo Comparator): Placebo (100% lactose) matched oral capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron — 8mg per day oral capsule
  Arms: Ondansetron
Drug: Placebo — daily oral capsule matched to active study medication. Made form 100% lactose powder
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the overall effectiveness of Ondansetron as an adjunctive or "add-on" medication in the treatment of Schizophrenia. This study is a double blind, placebo-controlled, randomised, 12 week trial.

DETAILED DESCRIPTION:
Ondansetron is a medication currently approved by the Australian Therapeutic Goods Administration for the treatment of drug-induced vomiting and nausea. Beyond this traditional use there have been several case reports and small clinical trials advocating the use of Ondansetron in the treatment of adult Schizophrenia. Overall these studies lend support to the use of Ondansetron in conjunction with mainstream antipsychotic medication in improving not only the positive symptoms associated with Schizophrenia but also the 'hard to treat' negative and cognitive symptoms. Furthermore, Ondansetron may also have potential benefits in reducing the adverse motor effects (e.g. tremor, uncontrolled muscle movements) associated with the use of many antipsychotic medications.

60 participants aged 18-65 inclusive with a DSM-IV diagnosis of Schizophrenia, Schizoaffective, or Schizophreniform disorder will be recruited. This study proposes to conduct a randomized, controlled treatment trial to investigate the efficacy of ondansetron as an adjunctive treatment in reducing negative and positive symptoms plus improving cognitive symptoms. There will be an initial screening session to determine participant suitability, a baseline session where the study medication (Ondansetron or Placebo) will be dispensed, followed by three monitoring visits.

The efficacy of Ondansetron will be evaluated by the following instruments:

* Positive and Negative Symptom Scale (PANSS)
* Montgomery-Åsberg Depression Rating Scale (MADRS)
* C-Reactive protein (marker of systematic and brain specific inflammation)

Safety will be assessed through adverse event reporting using the Adverse symptom Checklist (ASC), blood analysis, urinalysis, a 12-lead Electrocardiogram (ECG) and a physical examination. Adverse motor symptoms will also be assessed by the Abnormal Involuntary Movement Scale and the Simpson-Angus Scale. In addition a safety and monitoring committee consisting of research and medical staff external to the project will regularly review adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18-65 years of age
2. Have a current DSM-IV-TR diagnosis of schizophrenia, schizoaffective of schizophreniform disorders (diagnosis will be confirmed using the MINI Neuropsychiatric Interview)
3. Have been treated with a stable and standard dose (as determined by the PORT Treatment Recommendations for schizophrenia [33]) of an atypical antipsychotic agent (not including amisulpride owing to its 5HT3 actions) as their primary antipsychotic treatment for a minimum of eight weeks before entry into the trial
4. Are experiencing positive symptoms as evidenced by a score of >15 on the Positive Syndrome Subscale of the PANSS, and/or negative psychotic symptoms as evidenced by a score of >15 on the Negative Syndrome Subscale of the PANSS and /or significant cognitive dysfunction, as evidenced by at least 15 on the cognitive subscale. The cognition subscale used in this study, which included items of G10, G11, G12, P2, N5, and N7 from the PANSS were generated from previous studies.
5. Have a level of understanding sufficient to provide informed consent and to communicate with the investigators, study coordinator, and site personnel.

Exclusion Criteria:

1. Have an unstable medical condition, neurological disorder or an unstable seizure disorder. Any clinical significant electrocardiogram (ECG) abnormality at screening, including sinus bradycardia (ersting heart rate <50 beats per minute), atrial fibrillation, 2nd or 3rd degree AV block (AVB), prolonged ATc (QTcF>450ms in males or >470ms in females) history of congenital long AT syndromes, or risk of Torsades de Pointes because of family history of sudden death.
2. Currently pregnant or breastfeeding
3. Have a current DSM-IV-TR diagnosis of substance abuse or dependence disorder, or another Axis I disorder
4. Regularly use of another 5HT3 antagonist such as metoclopramide, cocaine, tropisetron, granisetron, palonosetron

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-07; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Symptom Scale (PANSS) | At screening visit and at three monitoring visits (week 4, week 8, week 12)
  The PANSS is a widely used, drug-sensitive, valid and reliable measure of psychopathology in schizophrenia. The PANSS is a formal interview, from which 30 symptoms are rated along a 7 point scale that ranges from 1 (absent) to 7 (extreme psychopathology). Schizophrenia symptom severity will be assessed with the PANSS and monitored to determine change in total, positive, negative, cognitive or general psychopathology symptoms.

SECONDARY OUTCOMES:
The Montgomery Åsberg Depression Rating Scale (MADRS) | At baseline visit and at three monitoring visits (week 4, week 8, week 12)
  The MADRS is a 10 item semi-structured clinician-rated interview of depression where each item (depression symptom) is rated of a 7 point scale ranging from 0 to 6. The MADRS will be used to monitor the participant's experience of depressive symptoms and severity across the trial.
Blood Test= C-Reactive Protein (CRP) | Screening visit and monitoring visit (week 12)
  CRP to determine changes in baseline levels in systemic and central nervous system inflammation)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Jayashri Kulkarni, Principal Investigator — Monash Alfred Psychiatry Research Centre (MAPrc)
Locations (1):
- Monash Alfred Psychiatry Research Centre (MAPrc), Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kulkarni J, Thomas N, Hudaib AR, Gavrilidis E, Gurvich C. Ondansetron - a promising adjunctive treatment for persistent schizophrenia. J Psychopharmacol. 2018 Nov;32(11):1204-1211. doi: 10.1177/0269881118798608. Epub 2018 Oct 25. PMID 30359166
- See also: Monash Alfred Psychiatry Research Centre (MAPrc) website — http://www.maprc.org.au